CLINICAL TRIAL: NCT04294641
Title: A Study of Front Line Ibrutinib Without Corticosteroids for Newly Diagnosed Chronic Graft-versus-Host Disease
Brief Title: Front Line Ibrutinib Without Corticosteroids for Newly Diagnosed Chronic Graft-versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200058; 20-C-0058
Record Dates: First submitted 2020-03-03; First posted 2020-03-04 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic GVHD
Keywords: Immunosuppressive Therapy; Kinase Inhibitors; steroid pulses; Hematologic Malignancies; alloHSCT
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Hematologic Neoplasms | interventions — ibrutinib; Electrocardiography; Respiratory Function Tests; Tomography, X-Ray Computed; Prednisone; Voriconazole; posaconazole; Azithromycin; montelukast; Budesonide; Beclomethasone; Filgrastim; pegfilgrastim; Erythropoietin; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ibrutinib Without Corticosteroids (Experimental): Determine response rate via continuous daily dose by mouth to determine efficacy
  Interventions: Drug: Ibrutinib; Diagnostic Test: ECG; Diagnostic Test: PFT's; Diagnostic Test: CT; Drug: Steroid pulse (prednisone); Drug: Voriconazole; Drug: Posaconazole; Drug: Azithromycin; Drug: Montelukast; Drug: Budesonide; Drug: Beclomethasone; Other: Filgrastim; Other: Pegfilgrastim; Other: Erythropoietin; Other: Transfusions; Procedure: Oral/Skin biopsy

INTERVENTIONS:
Drug: Ibrutinib — 140 mg capsules for a dose of 420 mg daily by mouth for up to 12 months.
  Other Names: Imbruvica
Diagnostic Test: ECG — At screening.
  Other Names: Electrocardiogram
Diagnostic Test: PFT's — Participants should have PFTs if not performed ≤3 months prior to start of study treatment and Cycle 7, Day 1 (6 months).
  Optional at Cycle 12, Day 28 (12 months) and Cycle 24, Day 28 (24 months).
  Other Names: Pulmonary function tests
Diagnostic Test: CT — Non-contrast CT at baseline and later during the study if clinically indicated.
  Other Names: Computed tomography
Drug: Steroid pulse (prednisone) — 0.5-2mg/kg/day allowed for clinical disease stabilization during first 4 weeks after starting Ibrutinib.
  Other Names: Rayos; Prednisone Intensol; Deltasone
Drug: Voriconazole — At any dose.
  Other Names: Vfend; Vfend IV
Drug: Posaconazole — As clinically indicated. At doses less than or equal to suspension 200 mg twice a day (BID) if ibrutinib dose modified to 280 mg once daily.
  OR Posaconazole suspension 200 mg three times a day (TID) or 400 mg BID if Ibrutinib dose modified to 140 mg once daily.
  OR Posaconazole injection intravenous (IV) injection 300 mg once daily; or delayed-release capsules 300 mg once daily if Ibrutinib dose modified to 140 mg once daily..
  Other Names: Noxafil
Drug: Azithromycin — Treat or prevent bronchiolitis obliterans.
  Other Names: AzaSite; Zithromax; Zithromax Z-Pak
Drug: Montelukast — Treat or prevent bronchiolitis obliterans.
  Other Names: Singulair
Drug: Budesonide — Treat or prevent gastrointestinal acute graft-versus host disease (GvHD).
  Other Names: Entocort; Uceris; Rhinocort Allergy
Drug: Beclomethasone — Treat or prevent gastrointestinal acute graft-versus host disease (GvHD).
  Other Names: Beclometasone; beclomethasone dipropionate; Qvar
Other: Filgrastim — Neutrophil growth factor permitted per institutional policy
  Other Names: Neupogen
Other: Pegfilgrastim — Neutrophil growth factor permitted per institutional policy.
  Other Names: Neulasta
Other: Erythropoietin — Red cell growth factor permitted per institutional policy.
  Other Names: haematopoietin; haemopoietin
Other: Transfusions — According to institutional policy.
Procedure: Oral/Skin biopsy — Optional. Baseline, Cycle 7, Day 1 (6 months), Cycle 12, Day 28 (12 months) and Cycle 24, Day 28.

SUMMARY:
Background:

- Chronic Graft Versus Host Disease (cGVHD) can occur after a person has had a stem cell or bone marrow transplant. In cGVHD, the donor cells attack the recipient's body. Researchers want to see if a drug called ibrutinib can block one of the proteins that lead to the immune reaction that causes cGVHD.

Objective:

- To see if ibrutinib as a first-line treatment can help people with newly diagnosed cGVHD.

Eligibility:

- People age 18 and older with newly diagnosed moderate or severe cGVHD

Design:

* Participants will be screened with:
* Medical and medicine histories
* Physical exam and vital signs
* Electrocardiograms (to measure heart function)
* Assessment of their ability to perform daily activities
* Blood and urine tests
* Assessment of their general well-being.
* Participants will visit the Clinical Center every 2 weeks for the first 2 months. Then they will visit every 4 weeks.
* Participants will take ibrutinib by mouth once every day of every cycle. One cycle is 28 days. Treatment will last up to 2 years. Participants will keep a medicine diary.
* Participants will take tests to measure lung function. They may have computed tomography scans of their chest. They will complete questionnaires about their symptoms and how cGVHD is affecting their body and quality of life. They will repeat the screening tests.
* Participants may have optional blood tests and/or skin biopsies to better understand the drugs effect on the body.
* Participants will be contacted by phone 30 days after treatment ends. They will also be contacted once a year for 2 years to discuss how they are feeling and if they have taken any other medicines to treat cGVHD.

DETAILED DESCRIPTION:
Background:

* Chronic graft-versus-host disease (GvHD) is the leading cause of late morbidity and non-relapse mortality following allogeneic hematopoietic stem cell transplantation (alloHSCT), occurring in 40-60% long-term survivors.
* Chronic GvHD occurs due to the dysfunctional peripheral tolerance during post-transplant hematopoietic reconstitution that allows the development and persistence of alloreactive donor-derived T and B cells.
* Prednisone is the front-line therapy; however, about 50% of participants have steroid-refractory disease and there is no standard second-line therapy.
* The most attractive approach for controlling chronic GvHD would be early therapy intervention which could prevent the most severe and irreversible clinical manifestations.
* Anti-B-cell therapy delivered early in chronic GvHD could be effective and steroid-sparing.
* Ibrutinib, reversible small molecule inhibitor of Brutons tyrosine kinase, has been shown to be well-tolerated and effective in phase 1b/2 trial for steroid refractory chronic GvHD.

Objective:

-To evaluate efficacy of ibrutinib as a first-line treatment for persons with newly diagnosed chronic GvHD by measuring the overall response rate (complete response [CR] + partial response [PR]) at 6 months, according to the 2014 National Institutes of Health (NIH) Consensus Criteria

Eligibility:

* Newly diagnosed, moderate or severe chronic GvHD according to the 2014 NIH Consensus Criteria, requiring systemic immunosuppression
* Age greater than or equal to 18 years old
* Karnofsky performance status greater than or equal to 60%
* History of prior alloHSCT; any donors, conditioning regimens and graft sources are allowed
* Adequate cardiac, hepatic and other organ function
* Adequate laboratory parameters

Design:

* Multi-center, non-randomized, phase II study
* Two-stage design will be used to determine the overall response rate (CR + PR) at 6 months
* Continuous daily dose of ibrutinib 420 mg by mouth, with the potential for dose reductions to 280 mg and 140 mg
* The accrual ceiling will be set at 40 participants, allowing for a total of up to 28 evaluable subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Newly diagnosed moderate or severe chronic Graft versus Host Disease (GvHD) (according to the 2014 National Institutes of Health (NIH) Consensus Criteria, requiring systemic immunosuppression.
  2. History of prior allogeneic Hematopoietic Stem Cell Transplant (HSCT) (any donors, conditioning regimens and graft sources are allowed).
  3. Subjects may have ongoing acute GvHD features (e.g., erythematous rash, elevated liver enzymes, diarrhea) which are in the opinion of the investigator responding to therapy.
  4. Stable doses of other immunosuppressive medications (e.g., calcineurin inhibitors, mycophenolate mofetil, rapamune, etc.) with no dose increase in the 2 weeks prior to study treatment initiation. Doses may be adjusted for trough levels.
  5. Age greater than or equal to 18 years old.
  6. Karnofsky performance status greater than or equal to 60%.
  7. Laboratory parameters as defined below:

     * Serum creatinine less than or equal to 2.0 x upper limit of normal (ULN).
     * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x ULN (less than or equal to 5 x ULN if unequivocal liver GvHD).
     * Total bilirubin less than or equal to 3 x ULN.
     * Absolute neutrophil count greater than or equal to 1.0 x 10(9)/L (no growth factor support allowed).
     * Platelets > 50 x 10(9)/L (no transfusions allowed less than or equal to 7 days prior to enrollment).
  8. Ability to understand and willingness to sign a written informed consent form.
  9. The effects of ibrutinib on the developing fetus are unknown. For this reason and because tyrosine kinase inhibitors may be teratogenic, female subjects of childbearing potential and men must agree to use highly effective methods of birth control (hormonal or barrier method of birth control; abstinence) prior to study entry, during the period of therapy, and for 30 days after the last dose of study drug.

EXCLUSION CRITERIA:

1. Relapsed or progressive malignant disease (other than minimal residual disease).
2. History of other malignant diseases, including post-transplant lymphoproliferative disease, with the following exceptions:

   * Malignancy treated with curative intent and with no evidence of active disease present for more than 3 years prior to prior to study treatment initiation and felt to be at low risk for recurrence.
   * Adequately treated non-melanomatous skin cancer or lentigo malignant melanoma without current evidence of disease.
   * Adequately treated cervical carcinoma in situ without current evidence of disease.
3. Received previous systemic treatment for chronic GvHD other than less than or equal to 0.5 mg/kg/day of prednisone equivalent for more than 7 days. Subject may be on steroids that were used to treat acute GvHD and then developed chronic GvHD before completing a taper. At the time of enrollment, the dose should be less than or equal to 0.5 mg/kg/day of prednisone equivalent with no dose increase in the preceding 2 weeks before study treatment initiation.
4. Prior or current treatment with:

   * Ibrutinib since the time of transplant (participants may have received ibrutinib prior to transplant for indications other than chronic GvHD).
   * Extracorporeal photopheresis (ECP) for acute GvHD less than or equal to 2 weeks prior to study treatment initiation; including any treatment with ECP for chronic GvHD.
   * Rituximab or other anti-B cell specific antibodies less than or equal to 4 weeks prior to study treatment initiation.
   * Any systemic investigational agents less than or equal to 4 weeks prior to study treatment initiation.
5. Impaired cardiac function including any one of the following:

   * Myocardial infarction, unstable angina or acute coronary syndrome less than or equal to 6 months prior to study treatment initiation.
   * Class 3 or 4 congestive heart failure, uncontrolled arrhythmia or uncontrolled hypertension at any time.
6. Uncontrolled infections (including prior aspergillosis) not responsive to antibiotics, antiviral medicines, or antifungal medicines.
7. Known bleeding disorder or subjects who received a strong cytochrome P450 (CYP) 3A inhibitor less than or equal to 7 days prior to the first dose of ibrutinib or requirement for continuous treatment with a strong CYP3A inhibitor.
8. Active hepatitis C virus (HCV) or hepatitis B virus (HBV). Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result to be enrolled.
9. Known hypersensitivity to ibrutinib.
10. Pregnant women are excluded from this study because ibrutinib has potential for teratogenic and abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ibrutinib, breastfeeding should be discontinued if the mother is treated with ibrutinib. Women who are planning to become pregnant and men who plan to father a child while enrolled in this study or less than or equal to 30 days after the last dose of study drug are excluded.
11. Any other reason at the discretion of the investigators and documented in the medical record that may raise concerns about the subject safety or ability to participate on this study.
12. Currently active, severe hepatic impairment Child-Pugh class C according to the Child Pugh classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Pavletic, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Washington University, School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-C-0058.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily: Ibrutinib Dose of 420 mg (3 x 140 mg capsules) daily by mouth for up to 12 months.
  Cohort 1: Participants with newly diagnosed moderate or severe chronic graft-versus-host disease) GvHD requiring systemic immunosuppression.
Period: Overall Study
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Started | 10
Completed | 6
Not Completed | 4
Not completed — Screen failure | 4

BASELINE CHARACTERISTICS:
Population: 4/10 participants were screen failures.
Groups:
- Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily: Ibrutinib Dose of 420 mg (3 x 140 mg capsules) daily by mouth for up to 12 months.
  Participants with newly diagnosed moderate or severe chronic graft-versus-host disease) GvHD requiring systemic immunosuppression.
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Baseline Global Scoring [Count of Participants; unit: Participants] — The global severity score is based on individual organ scores. Classifies chronic graft versus host disease participants as mild, moderate or severe based on the number of organs involved & the severity of disease in those organs. Each organ's severity is rated from 0 (no symptoms) - 3 (severe impairment/major disability). Mild: 1 or 2 organs involved with more than a score 1 plus lung score 0. Moderate: at least 1 organ (no lung) with a score of 2, OR- 3 or more organs involved with no more than score 1 OR lung score 1. Severe: at least 1 organ with a score of 3 OR lung score of 2 or 3.
  Participants
    Mild | 0
    Moderate | 3
    Severe | 3

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Participants With an Overall Response Rate (Complete Response [CR] + Partial Response [PR]) Reported With an 80% Confidence Interval at 6 Months
Description: To evaluate the efficacy of Ibrutinib as a first-line treatment for persons with newly diagnosed chronic graft-versus-host disease (GvHD) overall response rate was measured using the 2014 National Institutes of Health (NIH) consensus criteria and reported with an 80% confidence interval. CR is defined as complete resolution in all of signs and symptoms at all affected organs or tissues. PR is defined as improvement in ≥1 organ or tissue with no progression in any other affected organ or tissue.
Time Frame: At 6 months
Population: Six out of ten participants were analyzed because 4 participants were screen failures.
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Number analyzed (Participants) | 6
proportion of participants
  Complete Response | 0 [0 to 0.319]
  Partial Response | 0.1667 [0.0174 to 0.5103]

2. Primary Outcome: Fraction of Participants With an Overall Response Rate (Complete Response [CR] + Partial Response [PR]) Reported With an 95% Confidence Interval at 6 Months
Description: To evaluate the efficacy of Ibrutinib as a first-line treatment for persons with newly diagnosed chronic graft-versus-host disease (GvHD) overall response rate was measured using the 2014 National Institutes of Health (NIH) consensus criteria and reported with a 95% confidence interval. CR is defined as complete resolution in all of signs and symptoms at all affected organs or tissues. PR is defined as improvement in ≥1 organ or tissue with no progression in any other affected organ or tissue.
Time Frame: At 6 months
Population: Six out of ten participants were analyzed because 4 participants were screen failures.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Number analyzed (Participants) | 6
proportion of participants
  Complete Response | 0 [0.00 to 0.459]
  Partial Response | 0.167 [0.004 to 0.641]

3. Secondary Outcome: Fraction of Grade 3 and Grade 4 Serious and/or Non-serious Adverse Events in Participants With Newly Diagnosed Chronic Graft-versus-host Disease (GvHD)
Description: Safety of the agent will be determined by the fraction of grade of 3 and 4 serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 3 is severe, and Grade 4 is life-threatening.
Time Frame: Adverse events are captured from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the participant received the last study drug administration.
Population: Six out of ten participants were analyzed because 4 participants were screen failures.
Measure: Number (95% Confidence Interval); unit: proportion of adverse events
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Number analyzed (Participants) | 6
proportion of adverse events
  Grade 3 | 0.667 [0.223 to 0.957]
  Grade 4 | 0 [0.00 to -0.459]

4. Secondary Outcome: Failure-free Survival (FFS)
Description: Time to event endpoint failure free survival will be determined using a Kaplan-Meier curve and confidence intervals is calculated using the Brookmeyer-Crowley method. Failure-free survival (FFS) is defined as survival (from enrollment) without death, relapse of the underlying malignancy, or the addition of a new systemic chronic graft-versus-host-disease (GVHD) treatment.
Time Frame: Participants were followed from enrollment without death, relapse or new GVHD treatment up to 14 months
Population: Six out of ten participants were analyzed because 4 participants were screen failures.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Number analyzed (Participants) | 6
Months | 3.9 [2.5 to NA] — The upper confidence interval was not reached because limits are calculated using the Brookmeyer-Crowley method, and if the upper limit of the interval does not intersect the median, then it is recorded as not able to be estimated.

5. Secondary Outcome: Fraction of Participants Alive at 24 Months Follow-up Post-treatment
Description: Survival will be determined using a Kaplan-Meier curve at 24 months.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Number analyzed (Participants) | 6
proportion of participants | NA [NA to NA] — FFS at 24 months is reported as NA since no one's time from post treatment to death or last follow-up equals or exceeds 24 months.

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events are collected from the first study intervention, Study Day 1 of Cycle 1 through 30 days after the participant received the last study drug administration.
Population: Six out of ten participants were analyzed because 3 participants were screen failures, and one participant was ineligible.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: Beyond 30 days after the last intervention, only adverse events which are serious and related to the study intervention need to be recorded, up to 25 months.
Description: Six out of ten participants were analyzed because 4 participants were screen failures.
Arm/Group | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily
All-Cause Mortality (participants affected / at risk) | 3/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily (N=6)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 Ibrutinib Dose of 420 mg (3 x 140 mg Capsules) Daily (N=6)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 3 (4)
Fever (General disorders) | 1 (1)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastrointestinal disorders - Other, Soft stool (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Injury, poisoning and procedural complications - Other, Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Lymphocyte count increased (Investigations) | 1 (2)
Malaise (General disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 2 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — palpable superficial small cyst, patient reported it comes and goes, continue to monitor
Neutrophil count decreased (Investigations) | 2 (2)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT04294641/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/41/NCT04294641/ICF_001.pdf